CLINICAL TRIAL: NCT02157857
Title: A Molecular Test for Rapid On-site Evaluation in EBUS-TBNAsamples of Lung Cancer Patients
Brief Title: One Step Nucleic Acid Amplification in Endobronchial Ultrasound-guided Needle Aspiration Samples
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Filiz Oezkan, Dr. med. Filiz Oezkan, University Hospital, Essen
Other Study IDs: OSNA in EBUS-TBNA
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Lung Neoplasms
Keywords: NSCLC, SCLC, lung cancer, EBUS-TBNA
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Endobronchial ultrasound-guided needle-aspiration samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of our study is to investigate if CK19 mRNA-detection via OSNA can accurately detect lymph node metastases in lung cancer patients using EBUS-TBNA samples.

DETAILED DESCRIPTION:
Regional lymph nodes are assessed before tumor resection and before initiation of chemo- or radiotherapy. Endobronchial ultrasound-guided needle aspiration (EBUS-TBNA) is a well-established method for mediastinal and hilar lymph node staging [2, 3]. Samples obtained via this route are much smaller than surgical lymph node biopsies, yet they are able to provide complete and thorough evaluation, this includes current molecular testing.

One Step Nucleic Acid Amplification (OSNA), a molecular test that utilizes CK 19 mRNA-concentration as a target marker is becoming a rapidly dynamic method in quick detection of sentinel lymph node (SLN) metastases in breast cancer, colon cancer and other cancers.

In lung cancer, the role of SLN is not well established. However, recent publications suggest an accurate and rapid detection of lymph node metastases in NSCLC. However this requires complete lymph node dissection either with mediastinoscopy or by other surgical means such as thoracotomy.

The aim of our study is to investigate if CK19 mRNA-detection via OSNA can accurately detect lymph node metastases in lung cancer patients using EBUS-TBNA samples.

ELIGIBILITY:
Inclusion Criteria:

* CT-scan suspicious for lung cancer,
* enlarged mediastinal lymph nodes (>10 mm),
* EBUS-TBNA to be performed,
* age: 18-99 years

Exclusion Criteria:

* age: <18 years

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CT-scans suspicious for primary diagnosis of lung cancer and enlarged mediastinal lymph nodes Patients with known diagnosis of lung cancer and newly enlarged mediastinal lymph nodes
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-06 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
One step nucleic acid amplification of Cytokeratin 19 mRNA | 6 months
  One step nucleic acid amplification of Cytokeratin 19 mRNA, copy number detection

CONTACTS AND LOCATIONS:
Overall Officials: Kaid Darwiche, MD, Study Director — University Hospital, Essen; Filiz Oezkan, MD, Principal Investigator — University Hospital, Essen
Locations (1):
- Ruhrlandklinik, Essen, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Yasufuku K, Pierre A, Darling G, de Perrot M, Waddell T, Johnston M, da Cunha Santos G, Geddie W, Boerner S, Le LW, Keshavjee S. A prospective controlled trial of endobronchial ultrasound-guided transbronchial needle aspiration compared with mediastinoscopy for mediastinal lymph node staging of lung cancer. J Thorac Cardiovasc Surg. 2011 Dec;142(6):1393-400.e1. doi: 10.1016/j.jtcvs.2011.08.037. Epub 2011 Oct 2. PMID 21963329
- [Background] Inoue M, Hiyama K, Nakabayashi K, Morii E, Minami M, Sawabata N, Shintani Y, Nakagiri T, Susaki Y, Maeda J, Higashiyama M, Okami J, Yoshida Y, Ding J, Otomo Y, Okumura M. An accurate and rapid detection of lymph node metastasis in non-small cell lung cancer patients based on one-step nucleic acid amplification assay. Lung Cancer. 2012 Dec;78(3):212-8. doi: 10.1016/j.lungcan.2012.08.018. Epub 2012 Sep 29. PMID 23026640
- [Background] Babar M, Madani R, Thwaites L, Jackson PA, Devalia HL, Chakravorty A, Irvine TE, Layer GT, Kissin MW. A differential intra-operative molecular biological test for the detection of sentinel lymph node metastases in breast carcinoma. An extended experience from the first U.K. centre routinely offering the service in clinical practice. Eur J Surg Oncol. 2014 Mar;40(3):282-8. doi: 10.1016/j.ejso.2013.10.030. Epub 2013 Nov 21. PMID 24331309
- [Derived] Oezkan F, Khan AM, Hager T, Freitag L, Christoph D, Darwiche K. OSNA: A Fast Molecular Test Based on CK19 mRNA Concentration for Assessment of EBUS-TBNA Samples in Lung Cancer Patients. Clin Lung Cancer. 2016 May;17(3):198-204. doi: 10.1016/j.cllc.2015.09.001. Epub 2015 Sep 21. PMID 26455862